CLINICAL TRIAL: NCT06180343
Title: The Effect of Mandala Coloring on Students' Anxiety Level and Quality of Life
Acronym: Mandala
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Ayca Solt Kirca, Asssociate professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KırklareliAS-8
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Anxiety
Keywords: Mandala coloring; Stress
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomize controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala coloring group (Experimental): Participants will be asked to choose the pages they want from the 12 colored felt-tip pen paint sets and mandala coloring book given to each participant by the researcher, and color them in the colors they want, for 6 weeks, once a week, at any time of the day and for an average of 20-30 minutes each time.
  Participants will be asked to send a message before they start painting the mandala, and after the process, they will be asked to take a picture of the mandala they have painted and send it to the researcher. If the participants forget to color the mandala, a reminder message will be sent by the researcher twice a week.
  Interventions: Other: Mandala
- Control group (No Intervention): Participants in this group will consist of people who do not routinely do any practice on their own to reduce anxiety symptoms. Participants will be asked by telephone by the researcher twice a week for 6 weeks whether they have taken any action to reduce their anxiety symptoms. Participants who use any of the pharmacological or non-pharmacological practices to reduce anxiety symptoms will be excluded from the study.

INTERVENTIONS:
Other: Mandala — Participants will be asked to choose the pages they want from the 12 colored felt-tip pen paint sets and mandala coloring book given to each participant by the researcher, and color them in the colors they want, for 6 weeks, once a week, at any time of the day and for an average of 20-30 minutes each time.
  Participants will be asked to send a message before they start painting the mandala, and after the process, they will be asked to take a picture of the mandala they have painted and send it to the researcher. If the participants forget to color the mandala, a reminder message will be sent by the researcher twice a week.
  Arms: Mandala coloring group

SUMMARY:
Anxiety is a mood that focuses on the future, related to being prepared for possible upcoming negative events (fear, pain or danger), and unlike fear, its object is not determined or recognized, and it is exposed to uncertainty. Art therapy is used in the clinical and rehabilitation field as a useful tool for self-expression, healing and well-being. The close relationship between art, healing and well-being, and the therapeutic power of art has long been accepted all over the world.Many studies have been conducted in the literature examining the effect of mandala painting on reducing anxiety.This proposed project was planned to be carried out as a quasi-experimental study, based on the idea that mandala painting can reduce the level of anxiety in students and have a positive effect on the quality of life.

DETAILED DESCRIPTION:
Anxiety is a mood that focuses on the future, related to being prepared for possible upcoming negative events (fear, pain or danger), and unlike fear, its object is not determined or recognized, and it is exposed to uncertainty. Anxiety, which is felt as a common worry especially related to feelings of helplessness, is handled in two ways: state anxiety, which occurs in certain situations, and trait anxiety, which continues regardless of a specific situation.

Art therapy is used in the clinical and rehabilitation field as a useful tool for self-expression, healing and well-being. The close relationship between art, healing and well-being, and the therapeutic power of art has long been accepted all over the world. In line with developments in mental health since the mid-twentieth century, art has been widely appreciated as an important tool for both diagnosis and treatment. Art therapy offers individuals a safe haven to get away from past experiences and difficulties that no longer cause harm. In this context, there are many studies highlighting the effect of art therapy on psychological disorders such as healing trauma, death anxiety and burnout, showing that art therapy can be used as an alternative therapy in the treatment of emotion regulation and psychological disorders.

It is assumed that the repetitive patterns and symmetry of the mandala, which means circle in Sanskrit, create a meditative effect and increase psychological well-being by developing awareness. The anxiety-reducing effect of mandala, an integrative body-mind education form, has been associated with the circle; It is believed to increase psychological adaptation and preserve personality integrity, and is still used in psychotherapies today. Many studies have been conducted in the literature examining the effect of mandala painting on reducing anxiety.

When domestic and international literature is examined, it is noteworthy that there are no studies evaluating whether mandala painting reduces students' anxiety levels and increases their quality of life. This proposed project was planned to be carried out as a quasi-experimental study, based on the idea that mandala painting can reduce the level of anxiety in students and have a positive effect on the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Continuing her education at the Midwifery Department of the Faculty of Health Sciences
* Volunteering to participate in the study
* Knowing Turkish (being literate)

Exclusion Criteria:

* Having diagnosed psychiatric diseases,
* STAI anxiety score ≤36 (non-anxious)
* Having previously received non-pharmacological or pharmacological treatment

Ages: 19 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 60 (Estimated)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | 1 week
  The form consists of questions about socio-demographic

SECONDARY OUTCOMES:
World Health Organization Quality of Life Scale-Short Form (WHOQOL-BREF-TR) | 6 weeks
  The scale includes 27 questions in four areas: physical health, psychological health, social relations and environment. Questions are answered taking into account the last 15 days.
State-trait anxiety inventory | 6 weeks
  The State Anxiety Scale, which consists of twenty items, requires individuals to describe how they feel at a certain moment under certain conditions and to answer the items by taking into account their feelings about the situation. The total score obtained from the scale is between minimum 20 and maximum 80. Higher score it's mean worse.

CONTACTS AND LOCATIONS:
Overall Officials: AYCA SOLT KIRCA, Phd, Study Director — Kırklareli University

IPD SHARING:
Plan to Share IPD: No